CLINICAL TRIAL: NCT02851823
Title: Combined Application of ER:YAG and ND:YAG Lasers in Treatment of Chronic Periodontitis: A Split-mouth Randomized Controlled Trial
Brief Title: Combined Use of Er:YAG and Nd:YAG Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Dr. Mehmet Sağlam, Principal investigator, Department of Periodontology, Faculty of Dentistry, Izmir Katip Celebi University, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114S767
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Chronic Periodontitis
Keywords: Er-YAG lasers; Nd-YAG lasers; chronic periodontitis; nonsurgical periodontal debridement
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: split-mouth
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Control Group (Active Comparator): Mechanical periodontal treatment: Scaling and root planing were performed with periodontal curettes until the operator feels that root surface is clean, hard and smooth.
  Interventions: Device: Periodontal curettes
- Test Group (Experimental): Combined laser therapy: An Er:YAG laser (160 mj/pulse, 10 Hz) (AT Fidelis Fotona, Ljubljana, Slovenia) with water irrigation was first used to remove subgingival calculus and infected cementum.The Er:YAG laser beam was delivered into the periodontal pockets using a chisel-shaped quartz tip in contact mode under water irrigation, from a coronal to an apical direction with the tip inclined at 10o to 15o to the root surfaces. After Er:YAG laser application, Nd:YAG laser treatment (AT Fidelis Fotona, Ljubljana, Slovenia) was performed at an energy level of 100 mJ/pulse, and 20 Hz for removing pocket epithelium and detoxiﬁcation purpose. Irradiation was accomplished with a 320 μm fiber optic delivery system. The fiber was inserted into the periodontal pocket base in parallel alignment with the root surface, and the fiber was slowly moved from apical to coronal in a sweeping motion during the laser light emission.
  Interventions: Device: Er-YAG+Nd-YAG lasers

INTERVENTIONS:
Device: Periodontal curettes
  Other Names: Hu-Friedy, Gracey curets No. 1/2, 3/4, 5/6, 7/8, 11/12, 13/14, Hu-Friedy Ins. Co., USA
  Arms: Control Group
Device: Er-YAG+Nd-YAG lasers
  Other Names: AT Fidelis Fotona, Ljubljana, Slovenia
  Arms: Test Group

SUMMARY:
The aim of the present study was to compare the effectiveness of combined Er:YAG and Nd:YAG laser therapy to that of scaling and root planning with hand instruments in nonsurgical treatment of chronic periodontitis.

DETAILED DESCRIPTION:
The aim of the present study was to compare the effectiveness of combined Er:YAG and Nd:YAG laser therapy to that of scaling and root planning with hand instruments in nonsurgical treatment of chronic periodontitis.Twenty-ﬁve systemically healthy patients with moderate-to-advanced periodontal destruction were selected for this study. The quadrants were randomly allocated in a split-mouth design to either combined Er:YAG (160 mj/pulse, and 10 Hz) and Nd:YAG laser (100 mJ/pulse, and 20 Hz) therapy (test group) or scaling root planning using hand instruments (control group). At baseline, 1 month, and 3 months after treatment, clinical measurements, including plaque index (PI), gingival index (GI), probing depth (PD), clinical attachment level (CAL), and bleeding on probing (%) (BOP), were performed and gingival crevicular fluid and subgingival plaque samples were taken. The gingival crevicular fluid levels of interleukin-1β (IL-1β) and tumor necrosis factor-α (TNF-α) were analyzed by enzyme-linked immunosorbent assay. Total antioxidant status (TAS)/total oxidant status (TOS) were analyzed by high-performance liquid chromatography and a novel automatic colorimetric method. Quantitative analysis of Porphyromonas gingivalis (Pg), Tannerella forsythia (Tf), and Treponema denticola (Td) was performed using real-time polymerase chain reaction (PCR) procedures.

ELIGIBILITY:
Inclusion Criteria:

* The patients had ≥4 teeth per quadrant with probing depth (PD) of ≥5 mm, clinical attachment level (CAL) of ≥4 mm, and radiographic signs of alveolar bone loss. These individuals also had bleeding on probing (BOP) at >80% of the proximal sites.

Exclusion Criteria:

* Periodontal treatment received for the last 1 year; systemic diseases that could influence the outcome of the therapy, pregnancy, smoking, immunosuppressive chemotherapy; and use of antibiotics and anti-inflammatory drugs for the last 6 months.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Split-mouth design (test and control in the same patient).
Groups:
- Combined Er:YAG and Nd:YAG Laser vs Scaling and Root Planing: Combined Er:YAG and Nd:YAG Laser Application Left Side, Scaling and Root Planning Procedure Right Side" and "Scaling and Root Planning Procedure Left Side, Combined Er:YAG and Nd:YAG Laser Application Right Side
Period: Overall Study
Arm/Group | Combined Er:YAG and Nd:YAG Laser vs Scaling and Root Planing
Started | 25
1 Month (1 month after therapy) | 25
3 Months (3 months after therapy) | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Er:YAG+ Nd:YAG Laser Versus Scaling Root Planing: One side (left or right) of the mouth received Er:YAG+Nd:YAG laser therapy (test group) and other side received scaling and root planing with hand instruments (control group)
Arm/Group | Combined Er:YAG+ Nd:YAG Laser Versus Scaling Root Planing
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 25

OUTCOME MEASURES:

1. Primary Outcome: Clinical Attachment Level Change for Moderately Deep Pockets (4 mm≤PD≤6 mm)
Description: Change in clinical attachment level for moderately deep pockets (4 mm≤PD≤6 mm) between baseline and 1 month Change in clinical attachment level for moderately deep pockets (4 mm≤PD≤6 mm) between baseline and 3 month
Time Frame: Baseline, 1 and 3 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Control Group: Mechanical periodontal treatment: Scaling and root planing were performed with periodontal curettes until the operator feels that root surface is clean, hard and smooth.
  Periodontal curettes
- Test Group: Combined laser therapy: An Er:YAG laser (160 mj/pulse, 10 Hz) (AT Fidelis Fotona, Ljubljana, Slovenia) with water irrigation was first used to remove subgingival calculus and infected cementum.The Er:YAG laser beam was delivered into the periodontal pockets using a chisel-shaped quartz tip in contact mode under water irrigation, from a coronal to an apical direction with the tip inclined at 10o to 15o to the root surfaces. After Er:YAG laser application, Nd:YAG laser treatment (AT Fidelis Fotona, Ljubljana, Slovenia) was performed at an energy level of 100 mJ/pulse, and 20 Hz for removing pocket epithelium and detoxiﬁcation purpose. Irradiation was accomplished with a 320 μm fiber optic delivery system. The fiber was inserted into the periodontal pocket base in parallel alignment with the root surface, and the fiber was slowly moved from apical to coronal in a sweeping motion during the laser light emission.
  Er-YAG+Nd-YAG lasers
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 25 | 25
mm
  Change in CAL at 1 month | 2.07 (0.99) | 2.12 (0.97)
  Change in CAL at 3 months | 2.06 (1.04) | 2.09 (1.07)

2. Primary Outcome: Clinical Attachment Level Change for Deep Pockets (7 mm≤PD)
Description: Change in clinical attachment level for deep pockets (7 mm≤PD) between baseline and 1 month.
  Change in clinical attachment level for deep pockets (7 mm≤PD) between baseline and 3 month.
Time Frame: Baseline, 1 and 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 25 | 25
mm
  Change in CAL at 1 month | 3.74 (1.35) | 4.23 (0.99)
  Change in CAL at 3 months | 3.98 (1.45) | 4.66 (0.93)

ADVERSE EVENTS:
Arm/Group | Control Group | Test Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No